CLINICAL TRIAL: NCT03503318
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Risperidone Extended-Release Injectable Suspension (TV-46000) for Subcutaneous Use as Maintenance Treatment in Adult and Adolescent Patients With Schizophrenia
Brief Title: Study to Evaluate TV-46000 as Maintenance Treatment in Adult and Adolescent Participants With Schizophrenia
Acronym: RISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV46000-CNS-30072; 2018-001619-65 (EudraCT Number)
Record Dates: First submitted 2018-04-09; First posted 2018-04-19 (Actual); Results first posted 2021-12-09 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive an SC injection of placebo matching to TV-46000 at baseline and every 4 weeks (q4w) thereafter. Participants will continue treatment until they experience a relapse event; meet 1 or more of the study discontinuation or withdrawal criteria; or remain relapse-free during the double-blind phase until the study is terminated.
  Interventions: Drug: Placebo
- TV-46000 q1m (Experimental): Participants will receive an SC injection of TV-46000 at baseline and q4w thereafter. The maximal dose for adult participants is comparable to an oral risperidone dose of 5 milligrams (mg)/day, and the maximal dose for adolescents is comparable to 4 mg/day. Participants will continue treatment until they experience a relapse event; meet 1 or more of the study discontinuation or withdrawal criteria; or remain relapse-free during the double-blind phase until the study is terminated.
  Interventions: Drug: TV-46000
- TV-46000 q2m (Experimental): Participants will receive an SC injection of TV-46000 at baseline and every 8 weeks (q8w) thereafter, and a placebo SC injection 4 weeks after baseline and q8w thereafter. The maximal dose for adult participants is comparable to an oral risperidone dose of 5 mg/day, and the maximal dose for adolescents is comparable to 4 mg/day. Participants will continue treatment until they experience a relapse event; meet 1 or more of the study discontinuation or withdrawal criteria; or remain relapse-free during the double-blind phase until the study is terminated.
  Interventions: Drug: TV-46000; Drug: Placebo

INTERVENTIONS:
Drug: TV-46000 — TV-46000 will be administered per dose and schedule specified in the arm.
  Other Names: Risperidone
  Arms: TV-46000 q1m; TV-46000 q2m
Drug: Placebo — Placebo matching to TV-46000 will be administered per schedule specified in the arm.
  Arms: Placebo; TV-46000 q2m

SUMMARY:
The purpose of the study is to evaluate the efficacy, safety, and tolerability of different dose regimens of TV-46000 administered subcutaneously (SC) as compared to placebo during maintenance treatment in adult and adolescent participants with schizophrenia. The study will include male and female participants, 13 to 65 years of age, who have a confirmed diagnosis of schizophrenia, are clinically stable, and are eligible for risperidone treatment

ELIGIBILITY:
Inclusion Criteria:

* The participant has a diagnosis of schizophrenia for >1 year and has had ≥1 episode of relapse in the last 24 months.
* The participant has been responsive to an antipsychotic treatment (other than clozapine) in the past year based on discussions with family members or healthcare professionals.
* The participant has a stable place of residence for the previous 3 months before screening, and changes in residence are not anticipated over the course of study participation.
* The participant has no significant life events that could affect study outcomes expected throughout the period of study participation.
* Women of childbearing potential and sexually-active female adolescents must agree not to try to become pregnant, and, unless they have exclusively same-sex partners, must agree to use a highly effective method of contraception, and agree to continue use of this method beginning 1 month before the first administration of study drugs and for the duration of the study and for 120 days after the last injection of study drug.
* The participant, if adult or adolescent male, is surgically sterile, or, if capable of producing offspring, or has exclusively same-sex partners or is currently using an approved method of birth control and agrees to the continued use of this method for the duration of the study (and for 120 days after the last dose of study drug). Male participants with sex partners who are women of childbearing potential must use condoms even if surgically sterile

  * Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* The participant has a current clinically significant Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) diagnosis other than schizophrenia, including schizoaffective disorder, major depressive disorder, bipolar disorder, delirium, dementia, or amnestic or other cognitive disorders, or borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorder.
* The participant is currently on clozapine or received electroconvulsive therapy in the last 12 months.
* The participant has a history of epilepsy or seizures, neuroleptic malignant syndrome, tardive dyskinesia, or other medical condition that would expose the participant to undue risk.
* The participant has a positive serology for human immunodeficiency virus (HIV)-1, HIV-2, hepatitis B surface antigen, and/or hepatitis C.
* The participant has current or history of known hypersensitivity to risperidone or any of the excipients of TV-46000 or the oral formulation of risperidone used in the stabilization phase.
* The participant has a substance use disorder, including alcohol and benzodiazepines but excluding nicotine and caffeine.
* The participant has previously participated in a Teva-sponsored clinical study with TV-46000.
* The participant is a pregnant or lactating female.
* The participant has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery).
* The participant has used an investigational drug within 3 months prior to screening or has participated in a non-drug clinical trial within 30 days prior to screening.

  * Additional criteria apply, please contact the investigator for more information

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (81):
- United States (73):
  - Teva Investigational Site 14769, Little Rock, Arkansas
  - Teva Investigational Site 14796, Rogers, Arkansas
  - Teva Investigational Site 14811, Anaheim, California
  - Teva Investigational Site 14794, Bellflower, California
  - Teva Investigational Site 14776, Colton, California
  - Teva Investigational Site 14767, Costa Mesa, California
  - Teva Investigational Site 14802, Costa Mesa, California
  - Teva Investigational Site 14773, Culver City, California
  - Teva Investigational Site 14835, Garden Grove, California
  - Teva Investigational Site 14774, Glendale, California
  - Teva Investigational Site 14817, La Habra, California
  - Teva Investigational Site 14771, Lemon Grove, California
  - Teva Investigational Site 14823, Long Beach, California
  - Teva Investigational Site 14816, Montclair, California
  - Teva Investigational Site 14803, Norwalk, California
  - Teva Investigational Site 14786, Oakland, California
  - Teva Investigational Site 14797, Oceanside, California
  - Teva Investigational Site 14827, Oceanside, California
  - Teva Investigational Site 14777, Orange, California
  - Teva Investigational Site 14815, Pico Rivera, California
  - Teva Investigational Site 14812, Riverside, California
  - Teva Investigational Site 14785, San Bernardino, California
  - Teva Investigational Site 14818, San Diego, California
  - Teva Investigational Site 14828, San Diego, California
  - Teva Investigational Site 14819, San Marcos, California
  - Teva Investigational Site 14779, Santa Ana, California
  - Teva Investigational Site 14788, Torrance, California
  - Teva Investigational Site 14768, Coral Gables, Florida
  - Teva Investigational Site 14783, Coral Gables, Florida
  - Teva Investigational Site 14836, Hallandale, Florida
  - Teva Investigational Site 14787, Hialeah, Florida
  - Teva Investigational Site 14814, Hialeah, Florida
  - Teva Investigational Site 14799, Lauderhill, Florida
  - Teva Investigational Site 14832, Miami, Florida
  - Teva Investigational Site 14810, North Miami, Florida
  - Teva Investigational Site 14831, Orange City, Florida
  - Teva Investigational Site 14806, Orlando, Florida
  - Teva Investigational Site 14837, Tampa, Florida
  - Teva Investigational Site 14824, Atlanta, Georgia
  - Teva Investigational Site 14834, Columbus, Georgia
  - Teva Investigational Site 14821, Decatur, Georgia
  - Teva Investigational Site 14770, Marietta, Georgia
  - Teva Investigational Site 14765, Chicago, Illinois
  - Teva Investigational Site 14829, Chicago, Illinois
  - Teva Investigational Site 14805, Hoffman Estates, Illinois
  - Teva Investigational Site 14825, Shreveport, Louisiana
  - Teva Investigational Site 14764, Glen Burnie, Maryland
  - Teva Investigational Site 14820, New Bedford, Massachusetts
  - Teva Investigational Site 14798, Saginaw, Michigan
  - Teva Investigational Site 14791, St Louis, Missouri
  - Teva Investigational Site 14813, St Louis, Missouri
  - Teva Investigational Site 14826, St Louis, Missouri
  - Teva Investigational Site 14790, St Louis, Missouri
  - Teva Investigational Site 14809, Las Vegas, Nevada
  - Teva Investigational Site 14792, Berlin, New Jersey
  - Teva Investigational Site 14830, Princeton, New Jersey
  - Teva Investigational Site 14772, Cedarhurst, New York
  - Teva Investigational Site 14804, New York, New York
  - Teva Investigational Site 14800, New York, New York
  - Teva Investigational Site 14784, New York, New York
  - Teva Investigational Site 14780, Staten Island, New York
  - Teva Investigational Site 14763, Cincinnati, Ohio
  - Teva Investigational Site 14782, Dayton, Ohio
  - Teva Investigational Site 14822, Oklahoma City, Oklahoma
  - Teva Investigational Site 14789, Allentown, Pennsylvania
  - Teva Investigational Site 14833, Norristown, Pennsylvania
  - Teva Investigational Site 14775, Scranton, Pennsylvania
  - Teva Investigational Site 14793, Thorndale, Pennsylvania
  - Teva Investigational Site 14778, Charleston, South Carolina
  - Teva Investigational Site 14781, Dallas, Texas
  - Teva Investigational Site 14766, Dallas, Texas
  - Teva Investigational Site 14801, Houston, Texas
  - Teva Investigational Site 14807, Irving, Texas
- Bulgaria (8):
  - Teva Investigational Site 59148, Burgas
  - Teva Investigational Site 59152, Kazanlak
  - Teva Investigational Site 59151, Lovech
  - Teva Investigational Site 59149, Novi Iskar
  - Teva Investigational Site 59144, Sofia
  - Teva Investigational Site 59154, Varna
  - Teva Investigational Site 59150, Varna
  - Teva Investigational Site 59146, Vratsa

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.)

REFERENCES:
- [Derived] Kane JM, Tohami O, Franzenburg KR, Suett M, Sharon N, Merenlender-Wagner A, Eshet R, Harary E, Correll CU. Effects of Long-Term Treatment with TV-46000 on Symptom Improvement Over Time in Stabilized Patients with Schizophrenia. CNS Drugs. 2025 Nov 21. doi: 10.1007/s40263-025-01240-1. Online ahead of print. PMID 41272239
- [Derived] Correll CU, Knebel H, Harary E, Eshet R, Tohami O, Suett M, Sharon N, Franzenburg KR, Kane JM. Safety Outcomes with the Long-Acting Subcutaneous Antipsychotic TV-46000 in Schizophrenia: A Post Hoc Analysis of Behavioral, Neuromotor, Endocrine, and Cardiometabolic Outcomes from Two Phase 3 Studies. CNS Drugs. 2025 Nov;39(11):1139-1156. doi: 10.1007/s40263-025-01197-1. Epub 2025 Jul 29. PMID 40730715
- [Derived] Kane JM, Harary E, Eshet R, Tohami O, Weiser M, Leucht S, Merenlender-Wagner A, Sharon N, Davis GL 3rd, Suett M, Franzenburg KR, Correll CU. Efficacy and safety of TV-46000, a long-acting, subcutaneous, injectable formulation of risperidone, for schizophrenia: a randomised clinical trial in the USA and Bulgaria. Lancet Psychiatry. 2023 Dec;10(12):934-943. doi: 10.1016/S2215-0366(23)00288-2. Epub 2023 Nov 2. PMID 37924833

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to receive TV-46000 once monthly (q1m) subcutaneous (SC) injections, TV-46000 once every 2 months (q2m) SC injections, or placebo q1m SC injections in a 1:1:1 ratio. Open-label oral risperidone (2 to 5 mg/day) was used to stabilize participants to the treatments (the dose was based on clinical judgment) before randomization.
Groups:
- Placebo: Participants received an SC injection of placebo matched to TV-46000 at baseline and every 4 weeks (q4w) thereafter. Participants continued treatment until they experienced a relapse event; met 1 or more of the study discontinuation or withdrawal criteria; or remained relapse-free during the double-blind phase until the study was terminated.
- TV-46000 q1m: Participants received an SC injection of TV-46000 at baseline and q4w thereafter. The maximal dose administered to adult participants was comparable to an oral risperidone dose of 5 mg/day, and the maximal dose administered to adolescents was comparable to 4 mg/day. Participants continued treatment until they experienced a relapse event; met 1 or more of the study discontinuation or withdrawal criteria; or remained relapse-free during the double-blind phase until the study was terminated.
- TV-46000 q2m: Participants received an SC injection of TV-46000 at baseline and every 8 weeks (q8w) thereafter, and a placebo SC injection 4 weeks after baseline and q8w thereafter. The maximal dose administered to adult participants was comparable to an oral risperidone dose of 5 mg/day, and the maximal dose administered to adolescents was comparable to 4 mg/day. Participants continued treatment until they experienced a relapse event; met 1 or more of the study discontinuation or withdrawal criteria; or remained relapse-free during the double-blind phase until the study was terminated.
Period: Overall Study
Arm/Group | Placebo | TV-46000 q1m | TV-46000 q2m
Started | 181 | 183 | 180
Received at Least 1 Dose of Study Drug | 179 | 183 | 180
Completed | 142 | 144 | 140
Not Completed | 39 | 39 | 40
Not completed — Death | 1 | 0 | 4
Not completed — Adverse Event | 3 | 4 | 2
Not completed — Withdrawal by Subject | 12 | 17 | 16
Not completed — Protocol Violation | 5 | 0 | 3
Not completed — Lost to Follow-up | 17 | 15 | 12
Not completed — Other than specified | 1 | 3 | 3

BASELINE CHARACTERISTICS:
Population: Extended intent-to-treat (eITT) analysis set included all participants (adults and adolescents) randomized to the double-blind maintenance stage treatment, regardless if they had received treatment or not.
Groups:
- Placebo: Participants received an SC injection of placebo matched to TV-46000 at baseline and q4w thereafter. Participants continued treatment until they experienced a relapse event; met 1 or more of the study discontinuation or withdrawal criteria; or remained relapse-free during the double-blind phase until the study was terminated.
- TV-46000 q2m: Participants received an SC injection of TV-46000 at baseline and q8w thereafter, and a placebo SC injection 4 weeks after baseline and q8w thereafter. The maximal dose administered to adult participants was comparable to an oral risperidone dose of 5 mg/day, and the maximal dose administered to adolescents was comparable to 4 mg/day. Participants continued treatment until they experienced a relapse event; met 1 or more of the study discontinuation or withdrawal criteria; or remained relapse-free during the double-blind phase until the study was terminated.
- Total: Total of all reporting groups
Arm/Group | Placebo | TV-46000 q1m | TV-46000 q2m | Total
Number analyzed (Participants) | 181 | 183 | 180 | 544
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (11.43) | 50.6 (10.30) | 48.1 (11.09) | 49.3 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 71 | 70 | 212
  Male | 110 | 112 | 110 | 332
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 39 | 36 | 117
  Not Hispanic or Latino | 139 | 144 | 144 | 427
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 68 | 72 | 66 | 206
  Race: Black or African American | 104 | 108 | 110 | 322
  Race: Asian | 4 | 1 | 2 | 7
  Race: Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Race: Not Reported | 2 | 1 | 0 | 3
  Race: Other | 2 | 0 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to Impending Relapse (Number of Participants With Impending Relapse) for Intent-to-treat [ITT] Analysis Set
Description: Relapse was defined as 1 or more of the following items: • Clinical Global Impression-Improvement (CGI-I) of ≥5, and - an increase of any of the 4 Positive and Negative Syndrome Scale (PANSS) items: conceptual disorganization, hallucinatory behavior, suspiciousness, and unusual thought content, to a score of >4 with an absolute increase of ≥2 on specific item since randomization, or - an increase in any of the 4 individual PANSS items to a score of >4 and an absolute increase of ≥4 on combined score of 4 items since randomization; • hospitalization due to worsening of psychotic symptoms; • Clinical Global Impression-Severity of Suicidality (CGI-SS) of 4 (severely suicidal) or 5 (attempted suicide) on Part 1 and/or 6 (much worse) or 7 (very much worse) on Part 2; • violent behavior resulting in clinically significant self-injury, injury to another person, or property damage. Data is presented as distribution of relapsing participants (number of participants with impending relapse).
Time Frame: From randomization up to 108 weeks
Population: Intent-to-treat (ITT) analysis set included adult participants randomized to the double-blind maintenance treatment, regardless if they had received treatment or not.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TV-46000 q1m | TV-46000 q2m
Number analyzed (Participants) | 181 | 183 | 179
Participants | 53 | 13 | 23
Statistical Analysis 1: Comparison: Placebo vs TV-46000 q1m; Analysis was performed using the stratified Cox proportional hazard model, with treatment (placebo, TV-46000 q1m and TV-46000 q2m or placebo and TV-46000 overall [including q1m and q2m]) as explanatory variable and sex-dose as a stratification factor, and the stratified log rank test p-value (sex-dose as a stratification factor) referred to (TV-46000/placebo) comparison; Test type: Other; p < 0.0001, Log Rank — Threshold for significance at 0.05 level; Hazard Ratio (HR) = 0.200, 95% CI 2-sided [0.109 to 0.367]
Statistical Analysis 2: Comparison: Placebo vs TV-46000 q2m; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Log Rank — Threshold for significance at 0.05 level; Hazard Ratio (HR) = 0.375, 95% CI 2-sided [0.227 to 0.618]

2. Secondary Outcome: Time to Impending Relapse (Number of Participants With Impending Relapse) for Extended ITT [eITT] Analysis Set
Description: Relapse was defined as 1 or more of the following items: • CGI-I of ≥5, and - an increase of any of the 4 PANSS items: conceptual disorganization, hallucinatory behavior, suspiciousness, and unusual thought content, to a score of >4 with an absolute increase of ≥2 on specific item since randomization, or - an increase in any of the 4 individual PANSS items to a score of >4 and an absolute increase of ≥4 on combined score of 4 items since randomization; • hospitalization due to worsening of psychotic symptoms; • CGI-SS of 4 (severely suicidal) or 5 (attempted suicide) on Part 1 and/or 6 (much worse) or 7 (very much worse) on Part 2; • violent behavior resulting in clinically significant self-injury, injury to another person, or property damage. Data is presented as distribution of relapsing participants (adults and adolescents) (number of participants with impending relapse).
Time Frame: From randomization up to 108 weeks
Population: eITT analysis set included all participants (adults and adolescents) randomized to the double-blind maintenance stage treatment, regardless if they had received treatment or not.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TV-46000 q1m | TV-46000 q2m
Number analyzed (Participants) | 181 | 183 | 180
Participants | 53 | 13 | 24

3. Secondary Outcome: Proportion of Participants With Impending Relapse
Description: Relapse was defined as 1 or more of the following items: • CGI-I of ≥5, and - an increase of any of the 4 PANSS items: conceptual disorganization, hallucinatory behavior, suspiciousness, and unusual thought content, to a score of >4 with an absolute increase of ≥2 on specific item since randomization, or - an increase in any of the 4 individual PANSS items to a score of >4 and an absolute increase of ≥4 on combined score of 4 items since randomization; • hospitalization due to worsening of psychotic symptoms; • CGI-SS of 4 (severely suicidal) or 5 (attempted suicide) on Part 1 and/or 6 (much worse) or 7 (very much worse) on Part 2; • violent behavior resulting in clinically significant self-injury, injury to another person, or property damage. Impending relapse rate at Week 24 was estimated using the Kaplan-Meier product estimate.
Time Frame: Week 24
Population: ITT analysis set included adult participants randomized to the double-blind maintenance treatment, regardless if they had received treatment or not.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Placebo | TV-46000 q1m | TV-46000 q2m
Number analyzed (Participants) | 181 | 183 | 179
proportion of participants | 0.28 [0.205 to 0.347] | 0.07 [0.03 to 0.109] | 0.11 [0.065 to 0.165]

4. Secondary Outcome: Number of Participants Who Maintain Stability at the Endpoint
Description: Stability is defined as meeting all of the following criteria for at least 4 consecutive weeks: outpatient status; PANSS total score ≤80; minimal presence of specific psychotic symptoms on the PANSS, as measured by a score of ≤4 on each of the following items: conceptual disorganization, suspiciousness, hallucinatory behavior, and unusual thought content; Clinical Global Impression of Severity (CGI-S) score ≤4 (moderately ill); and CGI-SS score ≤2 (mildly suicidal) on Part 1 and ≤5 (minimally worsened) on Part 2. The last valid participant assessment was used as the endpoint.
Time Frame: At the endpoint (up to 108 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TV-46000 q1m | TV-46000 q2m
Number analyzed (Participants) | 181 | 183 | 179
Participants | 110 | 159 | 143

5. Secondary Outcome: Number of Participants Achieving Remission at the Endpoint
Description: The remission was achieved for participants who did not relapse during the study and for over a period of at least 6 months preceding the endpoint, maintained scores of = 3 on each of the 8 specific PANSS items: P1 (delusions), G9 (unusual thought content), P3 (hallucinatory behavior), P2 (conceptual disorganization), G5 (mannerisms/posturing), N1 (blunted affect), N4 (social withdrawal), and N6 (lack of spontaneity). The last valid participant assessment was used as the endpoint.
Time Frame: At Endpoint (up to 108 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TV-46000 q1m | TV-46000 q2m
Number analyzed (Participants) | 181 | 183 | 179
Participants | 30 | 39 | 42

6. Secondary Outcome: Observed Rate of Impending Relapse (Number of Participants With Impending Relapse) at the Endpoint
Description: Relapse was defined as 1 or more of the following items: • CGI-I of ≥5, and - an increase of any of the 4 PANSS items: conceptual disorganization, hallucinatory behavior, suspiciousness, and unusual thought content, to a score of >4 with an absolute increase of ≥2 on specific item since randomization, or - an increase in any of the 4 individual PANSS items to a score of >4 and an absolute increase of ≥4 on combined score of 4 items since randomization; • hospitalization due to worsening of psychotic symptoms; • CGI-SS of 4 (severely suicidal) or 5 (attempted suicide) on Part 1 and/or 6 (much worse) or 7 (very much worse) on Part 2; • violent behavior resulting in clinically significant self-injury, injury to another person, or property damage. Observed rate of impending relapse was calculated as the number of participants who relapsed by endpoint divided by the number of participants in each treatment group, using the last valid participant assessment as the endpoint.
Time Frame: At the Endpoint (up to 108 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TV-46000 q1m | TV-46000 q2m
Number analyzed (Participants) | 181 | 183 | 179
Participants | 53 | 13 | 23

7. Secondary Outcome: Time to Impending Relapse (Number of Participants With Impending Relapse) in the Adolescent Participants
Description: Relapse was defined as 1 or more of the following items: • CGI-I of ≥5, and - an increase of any of the 4 PANSS items: conceptual disorganization, hallucinatory behavior, suspiciousness, and unusual thought content, to a score of >4 with an absolute increase of ≥2 on specific item since randomization, or - an increase in any of the 4 individual PANSS items to a score of >4 and an absolute increase of ≥4 on combined score of 4 items since randomization; • hospitalization due to worsening of psychotic symptoms; • CGI-SS of 4 (severely suicidal) or 5 (attempted suicide) on Part 1 and/or 6 (much worse) or 7 (very much worse) on Part 2; • violent behavior resulting in clinically significant self-injury, injury to another person, or property damage. Data is presented as distribution of relapsing participants (adolescents) (number of participants with impending relapse).
Time Frame: From randomization up to 108 weeks
Population: eITT analysis set included all participants (adults and adolescents) randomized to the double-blind maintenance stage treatment, regardless if they had received treatment or not. Here, 'Overall number of participants analyzed' signifies adolescent participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TV-46000 q1m | TV-46000 q2m
Number analyzed (Participants) | 0 | 0 | 1
Participants |  |  | 1

8. Secondary Outcome: Change From Baseline in Drug Attitudes Inventory 10-item Version (DAI-10) Total Score at the Endpoint and End of Treatment
Description: The DAI-10 is a 10-item questionnaire to assess 1) subjective experience of drug and 2) attitudes and beliefs toward neuroleptics which may influence compliance in schizophrenia participants. The DAI-10 contains 6 items (1, 3, 4, 7, 9, and 10) that a participant who was fully adherent to the prescribed medication answered as "True" and 4 items (2, 5, 6, and 8) that a participant who was fully adherent to the prescribed medication answered as "False." A correct answer was scored +1 and an incorrect answer was scored -1. The total score was the sum of pluses and minuses, which ranged from -10 to 10 in increments of 2. A positive total score indicated a positive subjective response (compliant) and a negative total score indicated a negative subjective response (non-compliance). Higher scores denoted better compliance. The last valid participant assessment was used as the endpoint.
Time Frame: Baseline, endpoint and end of treatment (up to Week 108)
Population: ITT analysis set included adult participants randomized to the double-blind maintenance treatment, regardless if they had received treatment or not. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure, 'Number analyzed' signifies participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TV-46000 q1m | TV-46000 q2m
Number analyzed (Participants) | 178 | 182 | 179
units on a scale
  Baseline | 6.1 (3.23) | 5.8 (3.63) | 5.7 (3.13)
  Change at the Endpoint: number analyzed (Participants) | 125 | 139 | 137
  Change at the Endpoint | -0.8 (3.88) | 0.1 (3.34) | -0.3 (3.65)
  Change at the End of Treatment: number analyzed (Participants) | 55 | 84 | 79
  Change at the End of Treatment | -0.9 (3.42) | 0.3 (2.84) | 0.3 (3.51)

9. Secondary Outcome: Change From Baseline in Schizophrenia Quality of Life Scale (SQLS) Total Score at the Endpoint and End of Treatment
Description: The SQLS comprises 33 items categorized in 2 domains: psychosocial feelings (20 items) and cognition and vitality (13 items). The items were scored on a 5-point scale (1 - never, 2 - rarely, 3 - sometimes, 4 - often, 5 - always). Individual domain and total scores were standardized by scoring algorithm to a 0 (best health status) to 100 (worst health status) scale, with higher scores indicating comparatively lower quality of life. The last valid participant assessment was used as the endpoint.
Time Frame: Baseline, endpoint and end of treatment (up to Week 108)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TV-46000 q1m | TV-46000 q2m
Number analyzed (Participants) | 178 | 182 | 179
units on a scale
  Baseline | 34.0 (16.06) | 33.1 (16.79) | 34.2 (15.70)
  Change at the Endpoint: number analyzed (Participants) | 158 | 172 | 163
  Change at the Endpoint | 0.9 (14.24) | -4.5 (14.31) | -4.1 (15.23)
  Change at the End of Treatment: number analyzed (Participants) | 55 | 85 | 79
  Change at the End of Treatment | -2.3 (13.26) | -7.2 (13.79) | -7.3 (12.30)

10. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were defined as AEs occurring after the first dose of the study drug until 120 days after the last dose of study drug. Serious AEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: From randomization up to 120 days after last dose of study drug (up to Week 125)
Population: Safety analysis set included all randomized participants who received ≥1 dose of study treatment or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TV-46000 q1m | TV-46000 q2m
Number analyzed (Participants) | 179 | 183 | 180
Participants | 92 | 111 | 121

11. Secondary Outcome: Change From Baseline in Total Abnormal Involuntary Movement Scale (AIMS) Score at the End of Treatment
Description: The AIMS is a 14-item scale that includes assessments of orofacial movements, extremity and truncal dyskinesia, examiner's judgment of global severity, subjective measures of awareness of movements and distress, and a yes/no assessment of problems concerning teeth and/or dentures. Total AIMS score is a sum of item 1 through 7. Items 1 through 7 include facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). Each item was rated on a 0 (no dyskinesia) to 4 (severe dyskinesia) scale. Total AIMS score for Items 1-7 ranged from 0 to 28; with higher scores indicating greater severity of the condition.
Time Frame: Baseline, end of treatment (up to 108 weeks)
Population: Safety analysis set included all randomized participants who received ≥1 dose of study treatment or placebo. Here, 'Number analyzed' signifies participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TV-46000 q1m | TV-46000 q2m
Number analyzed (Participants) | 179 | 183 | 180
units on a scale
  Baseline | 0.4 (1.30) | 0.5 (1.83) | 0.2 (0.79)
  Change at the End of Treatment: number analyzed (Participants) | 55 | 93 | 81
  Change at the End of Treatment | 0.0 (1.10) | 0.1 (0.62) | 0.1 (1.00)

12. Secondary Outcome: Change From Baseline in Simpson-Angus Scale (SAS) Mean Score at the End of Treatment
Description: The SAS is a 10-item instrument for the assessment of neuroleptic-induced parkinsonism. The items on the scale include measurements of hypokinesia, rigidity, glabellar reflex, tremor, and salivation. Each item was rated on a 5-point scale (0 [None/Normal] to 4 [Extreme/Severe]). The mean score was calculated by adding the individual item scores and dividing by 10. The total mean score ranged from 0-4, with a higher score indicating greater severity of symptoms.
Time Frame: Baseline, end of treatment (up to 108 weeks)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TV-46000 q1m | TV-46000 q2m
Number analyzed (Participants) | 179 | 183 | 180
units on a scale
  Baseline | 0.07 (0.137) | 0.09 (0.195) | 0.06 (0.134)
  Change at the End of Treatment: number analyzed (Participants) | 55 | 93 | 81
  Change at the End of Treatment | 0.04 (0.134) | 0.02 (0.211) | 0.00 (0.102)

13. Secondary Outcome: Change From Baseline in Total Barnes Akathisia Rating Scale (BARS) Score at the End of Treatment
Description: The BARS is an instrument that assesses the severity of drug-induced akathisia. The BARS includes 3 items for rating objective restless movements, subjective restlessness, and any subjective distress associated with akathisia that were scored on a 4-point scale of 0 (normal/no distress) to 3 (constant restlessness/severe distress). Total score was the sum of scores of each item and ranged from 0-9, with higher scores indicating greater severity of akathisia.
Time Frame: Baseline, end of treatment (up to 108 weeks)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TV-46000 q1m | TV-46000 q2m
Number analyzed (Participants) | 179 | 183 | 180
units on a scale
  Baseline | 0.2 (0.63) | 0.1 (0.39) | 0.2 (0.57)
  Change at the End of Treatment: number analyzed (Participants) | 55 | 93 | 81
  Change at the End of Treatment | -0.1 (0.56) | 0.0 (0.51) | -0.1 (0.56)

14. Secondary Outcome: Number of Participants Reporting Suicidal Behavior and Suicidal Ideation Using Columbia-Suicide Severity Rating Scale (C-SSRS) at Baseline and Post-Baseline
Description: The C-SSRS is a semi-structured interview that captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal behavior was defined as a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation was defined as a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation.
Time Frame: Baseline, post-baseline (up to 108 weeks)
Population: Safety analysis set included all randomized participants who received ≥1 dose of study treatment or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TV-46000 q1m | TV-46000 q2m
Number analyzed (Participants) | 179 | 183 | 180
Participants
  Baseline: Suicidal behavior | 0 | 0 | 3
  Baseline: Suicidal ideation | 6 | 5 | 7
  Post-baseline: Suicidal behavior | 3 | 1 | 1
  Post-baseline: Suicidal ideation | 12 | 7 | 12

15. Secondary Outcome: Change From Baseline in Calgary Depression Scale for Schizophrenia (CDSS) Score at the End of Treatment
Description: The CDSS is specifically designed to assess the level of depression separate from the positive, negative, and EPS in schizophrenia. This clinician-administered instrument consists of 9 items, each rated on a 4-point scale from 0 (absent) to 3 (severe) that were added together to form the total CDSS depression score of the participant. The total score ranged from 0-27, with higher scores indicating greater severity of the condition.
Time Frame: Baseline, end of treatment (up to 108 weeks)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TV-46000 q1m | TV-46000 q2m
Number analyzed (Participants) | 179 | 183 | 180
units on a scale
  Baseline | 1.6 (2.14) | 1.3 (1.92) | 1.5 (1.93)
  Change at the End of Treatment: number analyzed (Participants) | 55 | 93 | 81
  Change at the End of Treatment | -0.4 (2.72) | -0.3 (1.39) | -0.8 (2.24)

16. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity of Suicidality (CGI-SS) Score at the End of Treatment
Description: The CGI-SS scale provides an overall clinician-rated assessment of the risk of suicidality. The CGI-SS consists of a 5-point scale in Part 1 (the most severe level of suicidality experience) ranging from 1 (not at all suicidal) to 5 (attempted suicide) and a 7-point scale in Part 2 (change in participant suicidality) ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: Baseline, end of treatment (up to 108 weeks)
Population: Safety analysis set included all randomized participants who received ≥1 dose of study treatment or placebo. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure, 'Number analyzed' signifies participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TV-46000 q1m | TV-46000 q2m
Number analyzed (Participants) | 179 | 183 | 179
units on a scale
  The most severe level of suicidality experience at Baseline | 1.0 (0.00) | 1.0 (0.00) | 1.0 (0.00)
  Change in participant suicidality at the End of Treatment: number analyzed (Participants) | 55 | 93 | 81
  Change in participant suicidality at the End of Treatment | 4.0 (0.00) | 4.0 (0.00) | 4.0 (0.00)

17. Secondary Outcome: Plasma Concentration of Risperidone, 9-OH-risperidone, and Total Active Moiety (Sum of Risperidone and 9-OH-risperidone)
Time Frame: 1 hour prior to dosing at Baseline (Day 1) and at the end of treatment visit (up to 108 weeks)
Population: Pharmacokinetics (PK) analysis set included all randomized participants who received ≥1 dose of study treatment or placebo and who also had ≥1 plasma concentration measured. Here, 'Number analyzed' signifies participants evaluable for specified categories.
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Placebo | TV-46000 q1m | TV-46000 q2m
Number analyzed (Participants) | 178 | 178 | 177
ng/mL
  Risperidone at Baseline | 4.694 [0.050 to 58.376] | 6.452 [0.050 to 97.935] | 5.364 [0.05 to 125.524]
  Risperidone at the End of Treatment: number analyzed (Participants) | 52 | 87 | 79
  Risperidone at the End of Treatment | 1.323 [0.050 to 47.683] | 13.215 [0.050 to 136.184] | 8.838 [0.05 to 75.95]
  9-OH-Risperidone at Baseline | 14.965 [0.150 to 84.471] | 18.473 [0.15 to 105.26] | 15.187 [0.15 to 107.316]
  9-OH-Risperidone at the End of Treatment: number analyzed (Participants) | 52 | 87 | 79
  9-OH-Risperidone at the End of Treatment | 2.982 [0.150 to 40.730] | 26.202 [0.15 to 101.354] | 17.778 [0.15 to 88.333]
  Total Active Moiety at Baseline | 19.060 [0.050 to 95.595] | 24.200 [0.050 to 134.202] | 19.945 [0.05 to 172.763]
  Total Active Moiety at the End of Treatment: number analyzed (Participants) | 52 | 87 | 79
  Total Active Moiety at the End of Treatment | 4.078 [0.050 to 62.621] | 38.429 [0.050 to 159.498] | 25.947 [0.05 to 135.823]

ADVERSE EVENTS:
Time Frame: From randomization up to 120 days after last dose of study drug (up to Week 125)
Description: Safety analysis set included only the randomized participants who received ≥1 dose of study treatment or placebo. No study drug was administered during the open-label stabilization period. All treatment-emergent adverse events are presented.
Arm/Group | Placebo | TV-46000 q1m | TV-46000 q2m
All-Cause Mortality (participants affected / at risk) | 1/179 | 0/183 | 4/180
Serious Adverse Events (participants affected / at risk) | 14/179 | 8/183 | 10/180
Other Adverse Events (participants affected / at risk) | 35/179 | 49/183 | 48/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=179) | TV-46000 q1m (N=183) | TV-46000 q2m (N=180)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 0/71 (0) | 1/71 (1) | 0/70 (0) — This is a gender-specific AE that affects only female participants.
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1)
Psychotic symptom (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 4 (5) | 0 (0) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=179) | TV-46000 q1m (N=183) | TV-46000 q2m (N=180)
Injection site nodule (General disorders) | 6 (20) | 12 (29) | 13 (23)
Injection site pain (General disorders) | 11 (37) | 9 (13) | 12 (14)
Injection site pruritus (General disorders) | 4 (5) | 10 (17) | 7 (10)
Weight increased (Investigations) | 6 (6) | 10 (10) | 13 (14)
Headache (Nervous system disorders) | 10 (11) | 9 (10) | 11 (11)
Insomnia (Psychiatric disorders) | 10 (11) | 12 (13) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2020-04-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT03503318/Prot_002.pdf
  • Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT03503318/SAP_003.pdf